CLINICAL TRIAL: NCT01567046
Title: Observational - Potentially Actionable Mutations in Archived Non-Rhabdomyosarcoma Soft Tissue Sarcomas (NRSTS)
Brief Title: Studying Genes in Tissue Samples From Younger and Adolescent Patients With Soft Tissue Sarcomas
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B5; NCI-2012-00714 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-27; First posted 2012-03-30 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Alveolar Soft-part Sarcoma; Childhood Angiosarcoma; Childhood Desmoplastic Small Round Cell Tumor; Childhood Epithelioid Sarcoma; Childhood Fibrosarcoma; Childhood Leiomyosarcoma; Childhood Liposarcoma; Childhood Malignant Mesenchymoma; Childhood Neurofibrosarcoma; Childhood Synovial Sarcoma; Chordoma; Desmoid Tumor; Metastatic Childhood Soft Tissue Sarcoma; Nonmetastatic Childhood Soft Tissue Sarcoma; Recurrent Childhood Soft Tissue Sarcoma
MeSH Terms: conditions — Hemangiosarcoma; Desmoplastic Small Round Cell Tumor; Sarcoma; Fibrosarcoma; Liposarcoma; Malignant mesenchymal tumor; Chordoma; Desmoid Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Archived DNA tissue samples are analyzed for frequency of genetic mutations, including SNPs, SNVs, and small deletions and/or insertions, by PCR and mass spectometry (Sequenom MassARRAY). Results are then analyzed to determine whether specific mutations correlate with patient or disease features such as tumor stage, histological grade, or outcome.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies genes in tissue samples from younger and adolescent patients with soft tissue sarcomas. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer

DETAILED DESCRIPTION:
Study Subtype: Ancillary/Correlative Observational Study Model: Cohort Time Perspective: Retrospective Biospecimen Retention: Samples With DNA Biospecimen Description: Tissue Study Population Description: Existing NRSTS samples from the COG D9902/ARST0332 studies Sampling Method: Non-Probability Sample

OBJECTIVES:

I. To determine the frequency with which actionable mutations are found in archived non-rhabdomyosarcoma soft tissue sarcoma (NRSTS) tumor specimens using mass spectrometry (MS) analysis of tumor-derived deoxyribonucleic acid (DNA).

OUTLINE:

Archived DNA tissue samples are analyzed for frequency of genetic mutations, including single nucleotide polymorphisms (SNPs), single nucleotide variants (SNVs), and small deletions and/or insertions, by polymerase chain reaction (PCR) and mass spectometry (Sequenom MassARRAY). Results are then analyzed to determine whether specific mutations correlate with patient or disease features such as tumor stage, histological grade, or outcome.

ELIGIBILITY:
Inclusion Criteria:

* Archived non-rhabdomyosarcoma soft tissue sarcoma (NRSTS) tumor-derived DNA

  * Synovial sarcoma, malignant peripheral nerve sheath tumor (MPNST), soft tissue sarcoma not otherwise specified (NOS), or other less common pediatric NRSTS
  * Formalin-fixed, paraffin-embedded (FFPE) tissue from patients enrolled on:

    * COG-D9902 Soft Tissue Sarcoma (STS) Biology and Banking Protocol
    * COG-ARST0332 A Risk-Based Treatment for Pediatric NRSTS Study
* See Disease Characteristics

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Non-rhabdomyosarcoma soft tissue sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of individual mutated genes in patients with NRSTS | Up to 1 month
Genetic changes that are most common and likely to have the greatest therapeutic impact | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Steve Skapek, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States